CLINICAL TRIAL: NCT01108536
Title: Dynamic Management of Excess Residual Limb Pressure With New Smart Socket Technology/Intelligent Amputee Sockets Employing Real Time Advanced Photonic Sensors for Optimum Fit and Pressure Relief Through Active Controls/Intelligent Prosthetic Socket With Variable Volume and Elevated Vacuum Systems
Brief Title: Dynamic Management of Excess Residual Limb Pressure With New Smart Socket Technology/Intelligent Prosthetic Socket With Variable Volume and Elevated Vacuum Systems
Acronym: SMARTsocket-
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Yiorgos, Dr., University of Wisconsin, Milwaukee
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CPSHI/IRB 00002053
Record Dates: First submitted 2010-03-22; First posted 2010-04-22 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Amputation
Keywords: prosthetics; socket comfort; amputation stump; amputee rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- adaptive trans-tibial socket (Experimental): subjects are fitted with experimental sockets.
  Interventions: Device: adaptive prosthetic socket

INTERVENTIONS:
Device: adaptive prosthetic socket — trans tibial socket with actuator zones (inflatable fluid bladders)
  Other Names: SMART socket

SUMMARY:
This study centers around the imaging of internal structures of residual limb by means of modern radiographic imaging techniques (Dynamic Radiography-DRSA).

The purpose of our research is to further study the behavior of bones and soft tissue of the socket-stump interface during dynamic tasks such as walking or brisk walking. In the long term this research could prove a basis for improvements in the general design of sockets for the new generation of prosthetic devices.

DETAILED DESCRIPTION:
There is very little known about the dynamic conditions inside a prosthetic socket, despite several research efforts based on pressure sensors, static X-ray images and/or computer simulations (FEM). The man reason is the inability of current measuring devices to track with enough resolution the in-vivo high speed kinematics of the stump-socket interface. Socket manufacturing and rectification in the field still relies on the experience and skill of the technician and feedback from the patient. This results in considerable dissatisfaction among the users and poor quantification of the socket fitting problems.

For lower extremity amputees, a well-fitting socket is an important element for a successful rehabilitation. The socket provides the interface between the prosthesis and residual limb, which is designed to provide comfort, appropriate load transmission, and efficient movement control. Attaining these objectives is extremely challenging, with up to 55% of lower limb amputees reporting dissatisfaction with socket comfort, residual limb pain, and/or skin breakdown. In addition, current techniques used to produce sockets with suitable characteristics are labor and cost intensive, and depend on the work of skilled prosthetists that are relatively scarce compared to the number of amputees. Currently, there are more than 500,000 lower limb amputees in the U.S. alone, with 60,000 new ones every year. For upper extremity amputees the issues related to the efficiency of movement, load transmission and comfort become even more challenging due to the different nature of the associated motor skills and performing tasks. Similarly there are l7,350 annual upper limb amputations distal to elbow in individuals under 21 years of age in the US. In most developed countries there are 1.55 amputees per 1000 people. Most amputees wear a prosthesis for about 70 hr/week and use crutches or wheelchairs as alternative assistive devices when performing certain tasks. Current solutions do not meet the patient specific needs.

It is suggested that our findings can further the understanding of the effects of slippage or harmful relative motion between stump and socket. Eventually new - and scientific based - guidelines for the fitting of artificial limbs could be recommended.

ELIGIBILITY:
Inclusion Criteria:

* trans-tibial amputation, proficiency in prosthesis use

Exclusion Criteria:

* pregnancy, balance impairment, stump skin breakdown

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Change in skin/socket displacement with different prosthetic sockets | one (1) year -baseline end of first year i.e. end of 2010 - with measurements at sixth and twelveth month

CONTACTS AND LOCATIONS:
Overall Officials: George Papaioannou, Ph.D, Principal Investigator — SAVE LLC
Locations (3):
- United States (2):
  - George Papaioannou Ph.d, New York, New York
  - Safe Llc Move Center and Laboratories, Milwaukee, New York, Nicosia, Wisconsin
- SAFE LLC, Nicosia, Cyprus, Cyprus